CLINICAL TRIAL: NCT01215864
Title: A Multicenter Phase I Study of TCD-717 Given by 4-Hour Intravenous Infusion in Patients With Advanced Solid Tumors
Brief Title: Study of Intravenous TCD-717 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Traslational Cancer Drugs Pharma, SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T10-10646
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Advanced Solid Tumors
Keywords: metastatic tumors; refractory tumors; recurrent tumors
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms

ARMS (1):
- TCD-717 (Experimental)
  Interventions: Drug: TCD-717

INTERVENTIONS:
Drug: TCD-717 — Patients will receive TCD-717 at the following dose levels:
  2, 4, 7, 10, 14, 19, 25, 31, 39, 49 or 61 mg/m^2

SUMMARY:
This is a Phase I dose escalation study of TCD-717, a novel drug that is a specific inhibitor of the enzyme choline kinase alpha, in patients with advanced solid tumors. The objectives of this study are to evaluate the safety of the drug and to determine the maximum tolerated dose and appropriate dose for phase II studies. Secondary objectives are to measure the efficacy of TCD-717; and in a substudy to be conducted in the MTD confirmation cohort only, to evaluate the potential correlation between the levels of tumor choline and tumor response to the choline kinase alpha inhibitor, TCD-717, using magnetic resonance spectroscopy. Pharmacokinetics analysis will be performed on patients enrolled in the maximum tolerated dose confirmation cohort.

DETAILED DESCRIPTION:
TCD Pharma has developed TCD-717, a novel drug that is a specific inhibitor of the enzyme choline kinase alpha (ChoKα), involved in the synthesis of phosphatidylcholine, which constitutes the major phospholipid in eukaryotic cell membranes and has been described as a potent oncogen when overexpressed in human cells. TCD-717 will be evaluated in this Phase I, open-label, single arm study to be performed at multiple centers. TCD-717 will be administered as a 4 hour infusion on two separate days per 7-day period per 28-day cycle (8 administrations per cycle). Eligible patients must have confirmed, metastatic or recurrent/refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically-confirmed solid tumors, metastatic or recurrent and refractory after standard therapy for the disease or for which conventional therapy is not reliably effective or no effective therapy is available.
2. Where possible, it is recommended that a paraffin block of tumor tissue or slides containing sections of tumor tissue be available (a sample should be collected and stored appropriately for the potential evaluation of choline kinase alpha expression in tumor tissue at the end of the study).
3. Patients must be ≥ 18 years of age.
4. Patients must have an ECOG Performance Status of 0, 1 or 2 and an estimated life expectancy of ≥ 12 weeks.
5. Patients must have adequate clinical laboratory values (i.e., absolute neutrophil count ≥1.5x10^9/L, platelets ≥100x10^9/L, plasma creatinine <= 1.5 x upper limit of normal (ULN) for the institution or a calculated creatinine clearance (using Cockroft and Gault formula) of ≥ 60 mL/min/1.73 m^2; bilirubin < 1.5 x ULN, alanine transaminase (ALT) and aspartate transaminase (AST) < 2.5 x ULN or ≤ 5 x ULN with liver involvement.
6. Patients may have either measurable or non-measurable disease as defined by RECIST.
7. Patients must give signed informed consent prior to the start of any study specific procedures.
8. Female patients with reproductive potential must have a negative serum or urine pregnancy test.
9. Patients with reproductive potential and their partners must be using at least one form of contraception as approved by the Investigator prior to study entry.
10. Patients with central nervous system metastases may be included if they are stable without administration of steroids. Patients with unstable metastatic CNS disease are excluded.

Exclusion Criteria:

1. Patients will be excluded if they have received previous anti-cancer chemotherapy, immunotherapy, vaccines, monoclonal antibodies, anti-angiogenic therapy, radiotherapy or any other investigational therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to study entry. Patients receiving concurrent anticancer therapy or intending to receive this at any time during the study will be excluded.
2. Patients who have received extensive prior radiotherapy to more than 30% of bone marrow reserves, or prior bone marrow/stem cell transplantation at any time prior to the study.
3. Patients with any concomitant condition that could compromise the objectives of this study and the patient's compliance.
4. Patients with significant cardiac disease including heart failure that meets New York Heart Association (NYHA) class III and IV definitions, history of myocardial infarction within six months of study entry, uncontrolled dysrhythmias or poorly controlled angina, uncontrolled hypertension or elevated heart rate.
5. Patients with a history of serious ventricular arrhythmia (VT or VF), QTc >=450 msec for men and 470 msec for women (as indicated in the ECG taken in the pre-treatment evaluation), or left ventricular ejection fraction (LVEF)<=50% by MUGA or Echocardiogram performed at the pre-treatment evaluation.
6. Pregnant or lactating females.
7. Patients with clinically evident HIV, HBV or HCV infection.
8. Patients with a hematologic malignancy.
9. Patients with a documented or known bleeding disorder or who require anticoagulation treatment that increases international normalized ratio (INR) or activated partial thromboplastin time (aPTT) above the institutional upper limit of normal.
10. Patients with clinically significant retinal abnormalities as per the medical history or ophthalmologic findings in the pre-treatment evaluation (e.g., retinitis pigmentosa or macular degeneration).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Safety of TCD-717 given by 4-hour intravenous infusion | Duration of the study
  Patients will be monitored throughout the study for adverse events and dose limting toxicities.

SECONDARY OUTCOMES:
Antitumor activity of TCD-717 given by 4-hour intravenous infusion | Duration of study
  Efficacy of TCD-717 will be asessed by RECIST 1.1
MTD confirmation cohort only: Pharmacokinetics (PK) of TCD-717 given by 4-hour infusion | Day 1-28 of Cycle 1
  For patients enrolled in MTD confirmation cohort, PK (Cmax, Tmax, AUC) will be measured during Cycle 1
To evaluate the potential correlation between the levels of tumor choline and tumor response to the choline kinase alpha inhibitor TCD-717 using magnetic resonance spectroscopy (MRS) (Substudy, MTD confirmation cohort only). | First scan will be pre-treatment (within 2 wks prior to start of treatment), then on Cycle 1 Day 25, and then within 7 days after determining disease progression
  MTD confirmation cohort only

CONTACTS AND LOCATIONS:
Overall Officials: Julie R Brahmer, MD, Principal Investigator — Johns Hopkins University; Patricia LoRusso, DO, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan